CLINICAL TRIAL: NCT06222775
Title: Multicomponent Intervention on Lifestyle, Anthropometric Measurements, Glycemic Control and Quality of Life in Patients Obese People With Type II Diabetes
Acronym: Diabesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 39/2023
Record Dates: First submitted 2023-12-21; First posted 2024-01-25 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: prevention; clinical trial; obesity; Diabetes Mellitus, Type 2; Healthy Lifestyle
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group receive activities on diabetes and obesity by Primary Care professionals on a care routine
  Interventions: Behavioral: Control Intervention 1; Behavioral: Control Intervention 2; Behavioral: Control Intervention 3; Behavioral: Control Intervention 4
- Experimental group (Experimental): Experimental group receive multicomponent intervention based on:
  De Cos AI, Gutiérrez Medina S, Luca B, Galdón A, Simon Chacín J, De Mingo ML, et al. Recommendations for clinical practice in diabetes and obesity. The Madrid Agreements. Document agreed by the working groups of the scientific societies: SENDIMAD, SOMAMFYC, SEMG Madrid, SEMERGEN Madrid and RedGDPS. Nutr Hosp [Internet]. 2018;35(4):971-8. Disponible en: http://dx.doi.org/10.20960/nh.1646 Kojdamanian Favetto V. Guía NICE 2022: actualización en el manejo de la diabetes mellitus tipo 2 en personas adultas. Evid actual pract ambul [Internet]. 2022;25(2):e007015. Disponible en: http://dx.doi.org/10.51987/evidencia.v25i3.7015
  Interventions: Behavioral: Group session 1; Behavioral: Group session 2; Behavioral: Group session 3; Behavioral: Group session 4; Behavioral: Group session 5; Behavioral: Group session 6; Behavioral: Group session 7 to 8; Behavioral: Group session 9

INTERVENTIONS:
Behavioral: Group session 1 — This session will have 3 editions in which the 50 participants of the experimental group will be distributed, with about 16 to 17 participants per edition.
  Its objective is to know the group and their expectations, in addition to providing basic knowledge about diabetes and a healthy lifestyle.
  Arms: Experimental group
Behavioral: Group session 2 — The sessions for the 5 groups will take place within 2 weeks. Two weeks after the 1st session, the 2nd session-workshop will be scheduled with no more than 10 participants. For this, 5 groups will be made. An attempt will be made to ensure that the participants in the groups remain stable.
  Its objective is to pave the way for the change to a healthy eating lifestyle and provide patients with sufficient knowledge so that with theory they can prepare a daily group menu according to the caloric needs of each of the participants.
  Arms: Experimental group
Behavioral: Group session 3 — Its general objective is to motivate the change towards healthy eating. And the specific ones develop a weekly menu according to calorie needs.
  Arms: Experimental group
Behavioral: Group session 4 — Its general objective is to reinforce a healthy lifestyle-eating, and the specific ones are to learn to read labels, preparing a weekly menu in a group.
  Arms: Experimental group
Behavioral: Group session 5 — Its general objective is to reinforce lifestyle-physical activity. And the specific objectives are to recognize that it is a moderate physical activity and the goal to achieve of recommended physical activity per week and plan a week of physical activity.
  Arms: Experimental group
Behavioral: Group session 6 — Its general objective is to reinforce a lifestyle-healthy eating and physical activity. And the specific ones are to reinforce the concept of physical activity in diabetes, what to do with hypoglycemia and adjust diet and exercise to current weight and needs.
  Arms: Experimental group
Behavioral: Group session 7 to 8 — The objective will be to maintain a healthy lifestyle and adjust menus and physical activity to current caloric needs, in addition to sharing experiences.
  Arms: Experimental group
Behavioral: Group session 9 — In the final session, a certificate of adherence to healthy living will be delivered, reminding you to continue with the acquired habits and attend scheduled consultations and tests.
  The days of the sessions are indicative, but they must be held in the week when the specified period of time between session and session is met.
  Other Names: Final session
  Arms: Experimental group
Behavioral: Control Intervention 1 — They will be given written information about the convenience of moderate physical activity and they will be informed of the importance of following an appropriate diet for diabetes and we will encourage weight loss.
  Arms: Control group
Behavioral: Control Intervention 2 — Your controls will be carried out according to the usual diabetes protocol established in the individual scheduled diabetes consultation reviews.
  Arms: Control group
Behavioral: Control Intervention 3 — These patients will also be given a written document about living with diabetes, advice on physical activity, and a pre-established diet will be given according to the number of calories needed previously calculated
  Arms: Control group
Behavioral: Control Intervention 4 — In addition to verbal recommendations. This document will be made after the act of assigning the control or experimental group.
  Arms: Control group

SUMMARY:
The main objective of this study will be to evaluate the effectiveness of a multicomponent intervention on nutritional recommendations and physical activity on glycemic control in obese patients with Type II Diabetes (DM2) in three places at the Algodonera Health Center of the Care Management Integrated in Talavera de la Reina.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic process that is not only important for its incidence and prevalence, but also for its complications. DM is responsible for cardiovascular complications that have high and premature mortality and a significant impact on quality of life. Diet control is one of the most effective therapeutic measures at all stages of diabetes management. It is important to promote healthy eating patterns that increase the consumption of foods with high nutritional value, in appropriate proportions, to improve overall health.

The objective of this study will be to evaluate the effectiveness of a multicomponent intervention on nutritional recommendations and physical activity on glycemic control in obese patients with Type II Diabetes (DM2) in three places at the Algodonera Health Center of the Integrated Care Management. from Talavera de la Reina.

For this purpose, a clinical trial will be carried out with two parallel arms, random assignment and blind evaluation by third parties. The study will be carried out on obese patients with DM2 between 40 and 75 years old at the "Algodonera" Health Center of the Integrated Care Management of Talavera de la Reina over a period of 1 year, from the subject's admission to the hospital. study until the last follow-up evaluation at one year. Selected patients must have a Barthel index > 90 and must travel to the health center independently.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a known diagnosis of DM2.
* Obese patients with a BMI > 30.
* Patients with Barthel index > 90
* Possibility of walking to the Health Center.
* Know how to read and write
* That they agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients with Type I DM.
* Inability to perform physical exercise, defined as such, that appears in your current medical history or that your PCP considers.
* Patients with complete deafness.
* Patients with blindness.
* Moderate or severe cognitive impairment.
* Participation in another clinical trial.
* Pregnant or breastfeeding women
* Any condition, laboratory parameter or concomitant therapy that, in the opinion of the investigator, may be a risk to the potential participant or that participation in the study is not in the best interest of the patient.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 12 months after the start of the study
  We expect a difference in the mean glycated hemoglobin between the control group and the experimental group of 0.6 units 12 months after starting participation in the study.

SECONDARY OUTCOMES:
Lipid profile (HDL) | 12 months after the start of the study
  Lipid profile (HDL) measure by mg/dL
Lipid profile (LDL) | 12 months after the start of the study
  Lipid profile (LDL) measure by mg/dL
Triglycerides | 12 months after the start of the study
  Triglycerides measure by mg/dL
Glomerular filtration rate | 12 months after the start of the study
  Measured glomerular filtration rate by ml/min
Proteinuria | 12 months after the start of the study
  Measured renal function by mg/dL
Weight | 12 months after the start of the study
  Body Weight (kg)
Body Mass Index | 12 months after the start of the study
  Body Mass Index measure as body weight (kg) divided by height (m) squared
Circumference weist | 12 months after the start of the study
  Circumference weist measure by cm
IPAQ - International Physical Activity Questionnaire | 12 months after the start of the study
  Physical activity measure by IPAQ in metabolic equivalents of tasks (METs)
PREDIMED - Prevention with Mediterranean diet | 12 months after the start of the study
  PREDIMED questionnaire to assess the adherence to the Mediterranean diet. 0 being the minimum total score and 14 the maximum total score. Higher values represent a higher adherence to the Mediterranean diet
SDSCA - Summary of Diabetes Self-Care Activities measure | 12 months after the start of the study
  Measures levels of behavior related to self-care and compliance with activities recommended by the doctor in the last 7 days in 5 areas (diet, exercise, blood glucose control, foot care and smoking) whose average score ranges from 0 and 7 (higher scores indicate better results)
Quality of life - Euroqol-5D | 12 months after the start of the study
  Evaluate the impact on the quality of life in people who participate in this project
Mortality of related to cardiovascular events | 12 months after the start of the study
  Heart failure, ischemic heart disease, stroke, kidney failure collected as such in patients electronic medical record
Morbility of related to cardiovascular events | 12 months after the start of the study
  Heart failure, ischemic heart disease, stroke, peripheral arterial disease, kidney failure, diabetic retinopathy, diabetic neuropathy collected as such in patients electronic medical record
Changes in medication diabetes | 12 months after the start of the study
  For the control of diabetes Glinids. Sulfonylureas. IDPP4. GLP1. Basal Insuline Mix insuline ISGLT2. Acarbose. Metformine.
Changes in Medication high blood pressure | 12 months after the start of the study
  For the control of high blood pressure IECAS. ARAII. Beta blockers Calcium antagonists Alpha blockers Diuretics
Changes in Medication cholesterol | 12 months after the start of the study
  For the control of cholesterol Statins Fibrates Fibrates + statins

CONTACTS AND LOCATIONS:
Overall Officials: Maria Salobrar Labrador García, Medical, Principal Investigator — Gerencia de Atención Integrada de Talavera de la Reina
Locations (1):
- Gerencia de Atención Integrada de Talavera de la Reina Centro de Salud La Algodonera, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lecube A, Monereo S, Rubio MA, Martinez-de-Icaya P, Marti A, Salvador J, Masmiquel L, Goday A, Bellido D, Lurbe E, Garcia-Almeida JM, Tinahones FJ, Garcia-Luna PP, Palacio E, Gargallo M, Breton I, Morales-Conde S, Caixas A, Menendez E, Puig-Domingo M, Casanueva FF. Prevention, diagnosis, and treatment of obesity. 2016 position statement of the Spanish Society for the Study of Obesity. Endocrinol Diabetes Nutr. 2017 Mar;64 Suppl 1:15-22. doi: 10.1016/j.endonu.2016.07.002. Epub 2016 Aug 16. No abstract available. English, Spanish. PMID 27543006
- [Background] Diabetes [Internet]. Who.int. [citado el 8 de julio de 2023]. Disponible en: https://www.who.int/es/news-room/fact-sheets/detail/diabetes
- [Background] OECD (2019), The Heavy Burden of Obesity: The Economics of Prevention, OECD Health Policy Studies, OECD Publishing, Paris, https://doi.org/10.1787/67450d67-en.
- [Background] Ampudia-Blanco FJ, Mata M. Diabetes tipo 2 en Atención Primaria. Evidencia y práctica clínica. Euromedice Ed Médicas. 2015;39-45
- [Background] Soriguer F, Goday A, Bosch-Comas A, Bordiu E, Calle-Pascual A, Carmena R, Casamitjana R, Castano L, Castell C, Catala M, Delgado E, Franch J, Gaztambide S, Girbes J, Gomis R, Gutierrez G, Lopez-Alba A, Martinez-Larrad MT, Menendez E, Mora-Peces I, Ortega E, Pascual-Manich G, Rojo-Martinez G, Serrano-Rios M, Valdes S, Vazquez JA, Vendrell J. Prevalence of diabetes mellitus and impaired glucose regulation in Spain: the Di@bet.es Study. Diabetologia. 2012 Jan;55(1):88-93. doi: 10.1007/s00125-011-2336-9. Epub 2011 Oct 11. PMID 21987347
- [Background] Astrup A, Finer N. Redefining type 2 diabetes: 'diabesity' or 'obesity dependent diabetes mellitus'? Obes Rev. 2000 Oct;1(2):57-9. doi: 10.1046/j.1467-789x.2000.00013.x. PMID 12119987
- [Background] Brunton SA. Diabesity. Clin Diabetes. 2022 Fall;40(4):392-393. doi: 10.2337/cd22-0088. No abstract available. PMID 36385971
- [Background] Costo-Muriel C, Martín-Carmona J, Pérez-Belmonte LM. Complicaciones macrovasculares de la diabetes. Medicine [Internet]. 2020;13(16):891-9. Disponible en: http://dx.doi.org/10.1016/j.med.2020.09.011
- [Background] Evert AB, Dennison M, Gardner CD, Garvey WT, Lau KHK, MacLeod J, Mitri J, Pereira RF, Rawlings K, Robinson S, Saslow L, Uelmen S, Urbanski PB, Yancy WS Jr. Nutrition Therapy for Adults With Diabetes or Prediabetes: A Consensus Report. Diabetes Care. 2019 May;42(5):731-754. doi: 10.2337/dci19-0014. Epub 2019 Apr 18. No abstract available. PMID 31000505
- [Background] Pérez-Rodrigo C, Hervás Bárbara G, Gianzo Citores M, Aranceta-Bartrina J. Prevalencia de obesidad y factores de riesgo cardiovascular asociados en la población general española: estudio ENPE. Rev Esp Cardiol [Internet]. 2022;75(3):232-41. Disponible en: http://dx.doi.org/10.1016/j.recesp.2020.12.013
- [Background] Thom G, Messow CM, Leslie WS, Barnes AC, Brosnahan N, McCombie L, Al-Mrabeh A, Zhyzhneuskaya S, Welsh P, Sattar N, Taylor R, Lean MEJ. Predictors of type 2 diabetes remission in the Diabetes Remission Clinical Trial (DiRECT). Diabet Med. 2021 Aug;38(8):e14395. doi: 10.1111/dme.14395. Epub 2020 Sep 27. PMID 32870520
- [Background] Leslie WS, Ford I, Sattar N, Hollingsworth KG, Adamson A, Sniehotta FF, McCombie L, Brosnahan N, Ross H, Mathers JC, Peters C, Thom G, Barnes A, Kean S, McIlvenna Y, Rodrigues A, Rehackova L, Zhyzhneuskaya S, Taylor R, Lean ME. The Diabetes Remission Clinical Trial (DiRECT): protocol for a cluster randomised trial. BMC Fam Pract. 2016 Feb 16;17:20. doi: 10.1186/s12875-016-0406-2. PMID 26879684
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Brosnahan N, Leslie W, McCombie L, Barnes A, Thom G, McConnachie A, Messow CM, Sattar N, Taylor R, Lean MEJ. Brief formula low-energy-diet for relapse management during weight loss maintenance in the Diabetes Remission Clinical Trial (DiRECT). J Hum Nutr Diet. 2021 Jun;34(3):472-479. doi: 10.1111/jhn.12839. Epub 2021 Jan 6. PMID 33406285
- [Background] Riobo Servan P. Obesity and diabetes. Nutr Hosp. 2013 Sep;28 Suppl 5:138-43. doi: 10.3305/nh.2013.28.sup5.6929. PMID 24010754
- [Background] Ballesteros Pomar MD, Vilarrasa Garcia N, Rubio Herrera MA, Barahona MJ, Bueno M, Caixas A, Calanas Continente A, Ciudin A, Cordido F, de Hollanda A, Diaz MJ, Flores L, Garcia Luna PP, Garcia Perez-Sevillano F, Goday A, Lecube A, Lopez Gomez JJ, Minambres I, Morales Gorria MJ, Morinigo R, Nicolau J, Pellitero S, Salvador J, Valdes S, Breton Lesmes I. The SEEN comprehensive clinical survey of adult obesity: Executive summary. Endocrinol Diabetes Nutr (Engl Ed). 2021 Feb;68(2):130-136. doi: 10.1016/j.endinu.2020.05.003. Epub 2020 Sep 12. English, Spanish. PMID 32933882
- [Background] De Cos AI, Gutierrez Medina S, Luca B, Galdon A, Simon Chacin J, De Mingo ML, Trifu D, Artola S, Egocheaga I, Soriano T, Vazquez C. [Recommendations for clinical practice in diabetes and obesity. The Madrid Agreements. Document agreed by the working groups of the scientific societies: SENDIMAD, SOMAMFYC, SEMG Madrid, SEMERGEN Madrid and RedGDPS]. Nutr Hosp. 2018 Aug 2;35(4):971-978. doi: 10.20960/nh.1646. Spanish. PMID 30070890
- [Background] Kojdamanian Favetto V. Guía NICE 2022: actualización en el manejo de la diabetes mellitus tipo 2 en personas adultas. Evid actual pract ambul [Internet]. 2022;25(2):e007015. Disponible en: http://dx.doi.org/10.51987/evidencia.v25i3.7015
- [Background] Europa.eu. 2012 [citado el 31 de agosto de 2023]. Disponible en: https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-clinical-investigation-medicinal-products-treatment-prevention-diabetes-mellitus-revision_en.pdf
- [Background] FDA. [citado el 31 de agosto de 2023].Guidance for Industry. Type 2 diabetes mellitus: evaluating the safety of new drugs for improving glycemic control. Draft; March 2020. Disponible en: https://www.fda.gov/media/135936/download
- [Background] Gummesson A, Nyman E, Knutsson M, Karpefors M. Effect of weight reduction on glycated haemoglobin in weight loss trials in patients with type 2 diabetes. Diabetes Obes Metab. 2017 Sep;19(9):1295-1305. doi: 10.1111/dom.12971. Epub 2017 May 22. PMID 28417575
- [Background] Organización Panamericana de la Salud (2019) [citado el 31 de agosto de 2023]. HEARTS Paquete técnico para el manejo de las enfermedades cardiovasculares en la atención primaria de salud. Hábitos y estilos de vida saludables: asesoramiento para los pacientes. Washington, D.C.: 2019. Disponible en: https://iris.paho.org/handle/10665.2/50805
- [Background] Córdoba García R, Camarelles Guillem F, Muñoz Seco E, Gómez Puente JM, San José Arango J, Ramírez Manent JI, et al. Recomendaciones sobre el estilo de vida. Actualización PAPPS 2022. Aten Primaria [Internet]. 2022;54(102442):102442. Disponible en: http://dx.doi.org/10.1016/j.aprim.2022.102442
- [Background] Orozco-Beltrán D, Brotons Cuixart C, Banegas Banegas JR, Gil Guillén VF, Cebrián Cuenca AM, Martín Rioboó E, et al. Recomendaciones preventivas cardiovasculares. Actualización PAPPS 2022. Aten Primaria [Internet]. 2022;54(102444):102444. Disponible en: http://dx.doi.org/10.1016/j.aprim.2022.102444
- [Background] Carrera Y . Cuestionario Internacional de actividad física Revista Enfermería del Trabajo 2017; 7:I1(49-54)
- [Background] Sociedad española de nutrición parenteral y enteral. Reunión de consenso sobre la metodología de las encuestas alimentarias, tipificación de la actividad física y estilos de vida saludables. Nutrición Hospitalaria, Laguardia 2014Vol. 31. Suplemento 3. marzo 2015.Disponible en: https://www.fen.org.es/anibes/archivos/documentos/nutr_hosp_supl_v31_2015.pd
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Salas-Salvado J, Diaz-Lopez A, Ruiz-Canela M, Basora J, Fito M, Corella D, Serra-Majem L, Warnberg J, Romaguera D, Estruch R, Vidal J, Martinez JA, Aros F, Vazquez C, Ros E, Vioque J, Lopez-Miranda J, Bueno-Cavanillas A, Tur JA, Tinahones FJ, Martin V, Lapetra J, Pinto X, Daimiel L, Delgado-Rodriguez M, Matia P, Gomez-Gracia E, Diez-Espino J, Babio N, Castaner O, Sorli JV, Fiol M, Zulet MA, Bullo M, Goday A, Martinez-Gonzalez MA; PREDIMED-Plus investigators. Effect of a Lifestyle Intervention Program With Energy-Restricted Mediterranean Diet and Exercise on Weight Loss and Cardiovascular Risk Factors: One-Year Results of the PREDIMED-Plus Trial. Diabetes Care. 2019 May;42(5):777-788. doi: 10.2337/dc18-0836. Epub 2018 Nov 2. PMID 30389673
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Caro-Bautista J, Morilla-Herrera JC, Villa-Estrada F, Cuevas-Fernandez-Gallego M, Lupianez-Perez I, Morales-Asencio JM. [Spanish cultural adaptation and psychometric validation of the Summary of Diabetes Self-Care Activities measure (SDSCA) among persons with type 2 diabetes mellitus]. Aten Primaria. 2016 Aug-Sep;48(7):458-67. doi: 10.1016/j.aprim.2015.08.005. Epub 2015 Dec 24. Spanish. PMID 26724986
- [Background] Collado Mateo D, Garcia Gordillo MA, Olivares PR, Adsuar JC. NORMATIVE VALUES OF EQ-5D-5L FOR DIABETES PATIENTS FROM SPAIN. Nutr Hosp. 2015 Oct 1;32(4):1595-602. doi: 10.3305/nh.2015.32.4.9605. PMID 26545523
- [Background] Herdman M, Badia X, Berra S. [EuroQol-5D: a simple alternative for measuring health-related quality of life in primary care]. Aten Primaria. 2001 Oct 15;28(6):425-30. doi: 10.1016/s0212-6567(01)70406-4. No abstract available. Spanish. PMID 11602124
- [Background] Ferriz, R., Sicilia, Á., & Lirola, M. J. "Cuestionario de la motivación para adoptar un estilo de vida saludable": Adaptación del Treatment Self-Regulation Questionnaire [Motivation Questionnaire to Adopt a Healthy Lifestyle: Adaptation of the Treatment SelfRegulation Questionnaire]. Behavioral Psychology, 2017 25(1), 79-97.
- [Background] Rubiales E. Consumo Energético Basal, según Mifflin [Internet]. SAMIUC. 2018 [citado el 9 de julio de 2023]. Disponible en: https://www.samiuc.es/consumo-energeticobasal-segun-mifflin
- [Background] Thom G, Gerasimidis K, Rizou E, Alfheeaid H, Barwell N, Manthou E, Fatima S, Gill JMR, Lean MEJ, Malkova D. Validity of predictive equations to estimate RMR in females with varying BMI. J Nutr Sci. 2020 May 26;9:e17. doi: 10.1017/jns.2020.11. PMID 32595965
- [Background] Cancello R, Soranna D, Brunani A, Scacchi M, Tagliaferri A, Mai S, Marzullo P, Zambon A, Invitti C. Analysis of Predictive Equations for Estimating Resting Energy Expenditure in a Large Cohort of Morbidly Obese Patients. Front Endocrinol (Lausanne). 2018 Jul 25;9:367. doi: 10.3389/fendo.2018.00367. eCollection 2018. PMID 30090085
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509